CLINICAL TRIAL: NCT04170361
Title: The Effect of Incentive Spirometry Added to Routine Physiotherapy Program on Hemodynamic Responses and Hospital Stay in Patients With COPD Exacerbation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: bvumkaya02
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: COPD Exacerbation
Keywords: COPD; incentive spirometry; length of stay; hemodynamic responses
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Patients will be admitted to chest physiotherapy program including breathing exercises, modified postural drainage and percussion, lower-upper extremity mobilization exercises and posture exercises once a day during hospitalization.
  Interventions: Other: Conventional Chest Physiotherapy
- Training Group (Experimental): In addition to conventional chest physiotherapy program, patients in this group will also be taught to use Triflo ® and apply at two-hour intervals.
  Interventions: Other: Conventional Chest Physiotherapy; Other: Conventional Chest Physiotherapy+Incentive Spirometry

INTERVENTIONS:
Other: Conventional Chest Physiotherapy — All patients will be admitted to physiotherapy rehabilitation program including breathing exercises, modified postural drainage and percussion, lower-upper extremity mobilization exercises and posture exercises once a day during hospitalization. In addition, patients in the education group will be taught the use of Triflo ® and administered at two-hour intervals. The program will be started within the first 24 hours and blood pressure, heart rate, oxygen saturation and respiratory frequency will be recorded before and after the sessions. The values obtained from the second session of the patients will be included in the analysis.
Other: Conventional Chest Physiotherapy+Incentive Spirometry — All patients will be admitted to physiotherapy rehabilitation program including breathing exercises, modified postural drainage and percussion, lower-upper extremity mobilization exercises and posture exercises once a day during hospitalization. In addition, patients in the education group will be taught the use of Triflo ® and administered at two-hour intervals. The program will be started within the first 24 hours and blood pressure, heart rate, oxygen saturation and respiratory frequency will be recorded before and after the sessions. The values obtained from the second session of the patients will be included in the analysis.In addition, patients in the education group will be taught the use of Triflo ® and administered at two-hour intervals.
  Arms: Training Group

SUMMARY:
COPD; it is a common, preventable and treatable disease that is associated with increased chronic inflammatory responses in the airways and lungs against harmful gases and particles, and that it manages progressive airflow. The definition of exacerbation is defined as an acute onset with a change in where daily differences in the main symptoms occur and which may occur with the presence of drugs. The number of exacerbations in the course of the disease is between 1-3 years on average. Routine physiotherapy treatment in COPD exacerbation is expected to increase lung volume and effective removal of airway secretions. The concept of physiotherapy programs is vibration, thoracic expression exercise, positive expiratory pressure therapy and gait programs.

An incentive spirometer is a simple, inexpensive device to adjust lung tissue re-expansion by increasing lung volumes and diaphragmatic mobility, providing maximal inspiration with termination control without a resistive loading. In COPD patients, the use of incentive spirometry is to increase alveolar ventilation and oxygenation in lifestyle.

There are a limited number of studies in the literature regarding the results of the use of incentive spirometry in COPD patients. The results of postoperative results of incentive spirometry in COPD patients were tried and established on pulmonary complications, diseases, postoperative dyspnea perception and lifestyle. The importance of the investigator's research; this is the first study to evaluate hemodynamic responses and hospitalization plans of incentive spirometer and routine physiotherapy program in COPD exacerbations.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with COPD exacerbation
* Hemodynamically stable
* To be conscious and voluntarily agree to participate in the study

Exclusion Criteria:

* Existence of neurological, cardiovascular and musculoskeletal problems to prevent exercise
* Having chronic respiratory disease other than COPD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-22 (Actual)

PRIMARY OUTCOMES:
Oxygen saturation | 30 minutes
  The oxygen saturation response will be measured before and after physiotherapy program with pulse oximeter.
Heart rate | 30 minutes
  The hearth rate response will be measured before and after after physiotherapy program with pulse oximeter.
Systolic and diastolic blood pressure | 30 minutes
  Blood pressure will be measured before and after physiotherapy program with monometer from the arm
Respiratory rate | 30 minutes
  Blood pressure will be measured before and after physiotherapy program with observation
Forced Vital Capacity (FVC) | 30 minutes
  FVC will be measured using MIR brand SPIRODOC model portable spirometer and expressed as the percentage of the predicted value according to the guideline of European Respiratory Society (ERS)
Forced Expiratory Volume in 1 second (FEV1) | 30 minutes
  FEV1 will be measured using MIR brand SPIRODOC model portable spirometer and expressed as the percentage of the predicted value according to the guideline of European Respiratory Society (ERS)
Peak Expiratory Flow (PEF) | 30 minutes
  PEF will be measured using MIR brand SPIRODOC model portable spirometer and expressed as the percentage of the predicted value according to the guideline of European Respiratory Society (ERS)
Forced Expiratory Volume 25-75% | 30 minutes
  FEF 25-75% will be measured using MIR brand SPIRODOC model portable spirometer and expressed as the percentage of the predicted value according to the guideline of European Respiratory Society (ERS)

CONTACTS AND LOCATIONS:
Overall Officials: Meltem Kaya, PT, PhD(c), Principal Investigator — Bezmialem Vakif University
Locations (2):
- Turkey (Türkiye) (2):
  - Meltem Kaya, Istanbul
  - Bezmialem Vakif University, Department of Physiotheraphy and Rehabilitation, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided